CLINICAL TRIAL: NCT03585725
Title: A Pilot Investigator-Initiated Study of Ribavirin in Indolent Follicular Lymphoma and Mantle Cell Lymphoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1709018594
Record Dates: First submitted 2018-05-25; First posted 2018-07-13 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Follicular Lymphoma; Mantle Cell Lymphoma
Keywords: Ribavirin; Follicular Lymphoma; Mantle Cell Lymphoma; Lymphoma; Non-Hodgkin lymphoma; Indolent Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma; Lymphoma, Non-Hodgkin | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ribavirin (Experimental): Ribavirin 1000 mg will be administered orally twice daily continuously in 28 day cycles for up to 6 cycles.
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — Ribavirin is FDA-approved oral medication for antiviral indications. Ribavirin will be obtained commercially for this trial.
  Treatment will be administered on an outpatient basis. Ribavirin should be administered with food.
  Other Names: Virazole; Rebetol; Copegus

SUMMARY:
This is a A Pilot Investigator-Initiated Study of Ribavirin in Indolent Follicular Lymphoma and Mantle Cell Lymphoma

DETAILED DESCRIPTION:
This clinical trial is for men and women ages 18 and older with follicular lymphoma with detectable BCL2-t or mantle cell lymphoma with presence of cyclin D1 overexpression (can be newly diagnosed or relapsed). The objective of this study is to assess the possibility of treating follicular lymphoma and mantle cell lymphoma patients with ribavirin and using cell free DNA (cfDNA) for BCL2-t and cyclin D1 extracted from peripheral blood to measure treatment effect.

Clinical trials of ribavirin have been conducted in relapsed and refractory acute myeloid leukemia (AML). Ribavirin, an antiviral agent with established doses, has resulted in the regression of the tumor.

* Ribavirin 1000 mg will be administered orally twice daily continuously for 28-day cycles.
* Patients will be followed for up to 7 months.
* Will continue on treatment as long as they are responding to therapy and not experiencing unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed follicular lymphoma with detectable BCL2-t or mantle cell lymphoma with presence of cyclin D1 overexpression (can be newly diagnosed or relapsed)
* Measurable disease (At least one tumor mass > 1 cm in diameter)
* Low tumor burden:

  1. No individual masses larger than 6 cm in diameter
  2. No more than three masses larger than 3 cm in diameter
  3. No lymphoma-related symptoms
* The treating physician does not feel that treatment with chemotherapy is indicated
* ECOG performance status of 0-2
* Adequate bone marrow and end organ function:

  i. ANC≥1500/mm3, hemoglobin≥10 g/dL, platelet≥100/mm3 ii. CrCL≥50 mL/min by Cockcroff Gault calculation

Exclusion Criteria:

* Indication for treatment of lymphoma including large tumor burden or symptomatic disease
* Pregnancy or men whose female partners are pregnant
* Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* Significant or unstable cardiac disease
* Hemoglobinopathy (thalassemia or sickle cell disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Number of participants who receive treatment for at least 3 months, have peripheral blood samples collected at baseline and monthly while on treatment, and have levels of BCL-t or cyclin D1, respectively, obtained from their peripheral blood samples | 18 months
  Feasibility will be measured by the number of subjects who receive ribavirin for at least 3 months, have peripheral blood samples collected at baseline and monthly while on treatment, and have levels of BCL-t and cyclin D1, respectively, obtained from their peripheral blood samples. The intervention will be deemed feasible if all three criteria are met in 10 out of 15 subjects.

SECONDARY OUTCOMES:
Number of participants with treatment-related Serious Adverse Events as assessed by the CTCAE v4.0 | 18 months
  Tolerability of ribavirin in FL and MCL will be assessed by the number of Number of participants with treatment-related Serious Adverse Events as assessed by the CTCAE v4.0.
Number of participants who achieve a response to ribavirin treatment based on PET/CT or CT | 18 months
  Response rate will be assessed by the number of participants who achieve a response to ribavirin treatment based on PET/CT or CT at baseline and within 4 weeks after completion of treatment. International working group criteria will be used for response assessment based on imaging done at baseline and 2-4 weeks after completion of therapy. The total number of participants who achieve a response will be assessed after the last patient has their response assessed after completion of therapy.
Average change in BCL2-t or Cyclin D1 cfDNA levels | 18 months
  Correlatives will be assessed by the change in BCL2-t or Cyclin D1 cfDNA levels. This will be correlated with response rates based on imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rutherford, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No